CLINICAL TRIAL: NCT04142814
Title: Randomized Controlled Study on the Evaluation of the T-PEP Method Based on Positive Expiratory Pressure Versus Intrapulmonary Percussive Ventilation for Lower Respiratory Airways Clearance in Sub-acute, Tetraplegic, Tracheotomized Spinal Cord Injured Patients
Brief Title: Randomized Controlled Study on T-PEP Versus IPV Method for Lower Respiratory Airways Clearance in Tetraplegic Tracheotomized Spinal Cord Injured Patients
Acronym: T-PEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients case mix changed and did not match anymore with selection criteria
Sponsor: Montecatone Rehabilitation Institute S.p.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE-378/2018/SPER/AUSLIM
Record Dates: First submitted 2019-10-22; First posted 2019-10-29 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Spinal Cord Injury Cervical
Keywords: Lower respiratory airways clearance; Deep lung clearance; Secretions overproduction; Positive Expiratory Pressure; Intrapulmonary Percussive Ventilation; Tetraplegia; Tracheotomy; Critical Care Unit; Mechanical ventilation; Respiratory physiotherapy
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-PEP (Experimental): Each T-PEP session includes 10 inspiratory/expiratory cycles, repeated 3 times and interspersed by a pause of about 3 minutes.
  Each session will be immediately followed by bronchoaspiration and/or Mechanical Insufflation-Exsufflation (MI-E).
  Sessions will take place at least twice a day for a number of days until the attainment of an effective pulmonary ventilation (as detected by thoracic auscultation), then continued for a further 3 days (at least 2 times a day) for the outcome stabilization, as confirmed also by arterial-blood gas test (ABG), spirometry, chest X-ray and chest ultrasound.
  T-PEP sessions will take place at least 1 hour after meals or nutrition via nasogastric tube.
  Tracheal cannula will be kept constantly cuffed during the sessions. Ipratropium Bromide treatment will be on place from study entry until at least 4 weeks after the attainment of a stabilized effective pulmonary ventilation.
  Interventions: Procedure: T-PEP
- IPV (Active Comparator): Each IPV session includes 3 treatment cycles, interspersed with a pause, consisting of a first high-frequency steps, lasting about 5 minutes, immediately followed by a second low-frequency step lasting approximately one minute.
  Each session will be immediately followed by bronchoaspiration and/or Mechanical Insufflation-Exsufflation (MI-E).
  Sessions will take place at least twice a day for a number of days until the attainment of an effective pulmonary ventilation (by thoracic auscultation), then continued for a further 3 days (at least 2 times a day) for outcome stabilization, as confirmed by ABG test, spirometry, chest X-ray and chest ultrasound.
  IPV sessions will take place at least 1 hour after meals or nutrition via nasogastric tube.
  Tracheal cannula will be kept constantly cuffed during the sessions. Ipratropium Bromide treatment will be on place from study entry until at least 4 weeks, after the attainment of a stabilized effective pulmonary ventilation.
  Interventions: Procedure: IPV

INTERVENTIONS:
Procedure: T-PEP — First of all, a corrugated tube for ventilation is assembled: in one end with an antibacterial filter for ventilation and then an inflation system (like Auxiliary Manual Breathing Unit - AMBU); in the other end with a connector and then a one-way PEP Valve. The latter holds a junction for the tracheal cannula and a pressure gauge. A Venturi Resistor is placed in the expiratory part of the PEP Valve.
  After connection to the tracheal cannula, the disostructive maneuver is manually executed by a respiratory physiotherapist.
  Arms: T-PEP
Procedure: IPV — IPV is delivered via a commercial device that can be set by frequency, duration of inspiratory time, inspiratory-expiratory ratio and positive end-expiratory pressure, based on patients characteristics and clinical needs. It is connected to the patient's tracheal cannula via a Mount catheter. The air supplied is sterile, due to the presence of an antibacterial filter present in the device.
  Arms: IPV

SUMMARY:
In tetraplegic patients with complete cervical spinal cord injury, respiratory complications are very frequent, especially in the sub-acute phase: the lungs often become obstructed due to the accumulation of secretions and the contemporary inefficiency of the cough mechanism. The present pilot study aims, in the context of a rehabilitative Critical Care Unit, at evaluating a not yet published method, called "T-PEP" and based on the principle of Positive Expiratory Pressure, applicable to tracheotomised and mechanically ventilated patients. This method, conceptually simple and low cost, is compared with a known method based on the principle of Percussive Intrapulmonary Ventilation (IPV). Safety and efficacy issues are covered.

DETAILED DESCRIPTION:
Respiratory complications are very frequent, especially in the sub-acute phase following a spinal cord injury and must be treated to avoid even very serious outcomes. In the patient with a complete cervical spinal cord injury (and therefore tetraplegic, from a motor perspective), the lungs often become obstructed due to the accumulation of secretions and the contemporary inefficiency of the physiological mechanism of the cough. Various methods for bronchial clearance are known, but when the patient is tracheotomized and the secretions accumulate in the deepest part of the lung, nowadays the only described method available to mobilize such secretions and allow more efficient respiratory exchanges is based on the principle of Percussive Intrapulmonary Ventilation (IPV). It requires a special device, equipped with a pneumatic air generator, connected to the tracheal cannula. Such treatment needs the assistance of highly trained and expert operators, moreover IPV is a quite complex and expensive technique which has to be applied in a prudential manner in such tetraplegic patients, especially because they show significant hemodynamic instability in the acute/sub-acute phase after the spinal cord lesion.

The principle of Positive Expiratory Pressure (PEP) is already known for its efficacy in the secretions' clearance of the lower respiratory airways in other pathological conditions. However, in its classic modalities, it requires the preservation of the functionality of the respiratory muscles. To circumvent this limit in tetraplegic and tracheotomized patients, a respiratory physiotherapeutic procedure called "T-PEP" has been developed at the Montecatone Rehabilitation Institute. Such method is conceptually simple and low cost, it requires the manual assistance of a trained physiotherapist and the use of some components of common use in the clinical practice of Critical Care Units.

The present pilot randomized controlled trial aims at comparing the T-PEP and IPV methods, assigned to 2 parallel arms (1:1 allocation ratio), in the context of the Critical Care Unit of the Montecatone Rehabilitation Institute hospital, in sub-acute, tetraplegic, tracheotomized, mechanically ventilated, spinal cord injured patients. The trial covers safety and efficacy issues; cognitive performances are also addressed.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord injury due to traumatic or non-traumatic etiology;
* neurological level from C4 to C7 (included)
* complete spinal cord injury, classifiable as "A" grade according to the Asia Impairment Scale (AIS);
* distance from the spinal cord injury event from 1 to 5 weeks;
* first admission to Montecatone R.I. (in particular to the Critical Care Unit);
* patients with middle-basal hypoventilation;
* patients in partial or continuous mechanical ventilation;
* patients with tracheotomy;
* patients capable of giving meaningful consent;
* collaborating patients.

Exclusion Criteria:

* thoracic trauma with non-drained thoracic fractures and / or pneumothorax and / or hemorrhage;
* pleural effusion;
* significant hemodynamic instability needing amines administration and / or Shock Index > 1.5;
* patients with tracheoesophageal fistulae;
* patients with severe acquired brain injury;
* patients with ongoing sepsis;
* patients with ongoing pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Through the whole period of clearance treatment to attain a stabilized effective pulmonary ventilation (whole period length is 2 weeks on average) until the following 4 weeks
  Incidence of adverse events in the treatment period and during the subsequent follow-up, directly correlated with the lower airways cleaning treatments under investigation

SECONDARY OUTCOMES:
Time needed for attainment of a stabilized effective pulmonary ventilation | Through the whole period of clearance treatment to attain a stabilized effective pulmonary ventilation (whole period length is 2 weeks on average)
  Number of days needed to attain the stabilization of an effective pulmonary ventilation, as confirmed simultaneously by all the following examinations: chest auscultation, ABG (for respiratory exchanges efficiency), spirometry (in particular: Forced Expiratory Flow 75% [FEF 75], for pulmonary patency), chest X-ray and chest ultrasound.
Recurrence of lower airways obstruction | From the attainment of stabilized effective pulmonary ventilation until 3 months later
  Incidence of recurrence of lower airways obstructions requiring retreatment with the lower airways treatments under investigation, in the study period following the attainment of stabilized effective pulmonary ventilation
Incidence of infections of lower respiratory airways | Through the whole period of clearance treatment to attain a stabilized effective pulmonary ventilation (whole period length is 2 weeks on average) and through the following 3 months
  Incidence of acute infections of the lower respiratory airways, throughout the study period.
Incidence of sepsis | Through the whole period of clearance treatment to attain a stabilized effective pulmonary ventilation (whole period length is 2 weeks on average) and through the following 3 months
  Incidence of sepsis related to acute infections of the lower respiratory airways, throughout the study period
Time needed for weaning from mechanical ventilation, from its start | From mechanical ventilation start date until mechanical ventilation end date (up to 1 year)
  Number of days needed to wean from mechanical ventilation, starting from the mechanical ventilation starting date (also if previously occurred in a sending hospital)
Time needed for weaning from mechanical ventilation, from hospital admission | From admission date to Montecatone R.I. until mechanical ventilation end date (up to 1 year)
  Number of days needed to wean from mechanical ventilation, starting from the date of admission to the Montecatone R.I. hospital
Evaluation of cognitive performance: attention and memory - 1 | Baseline (initial visit); day of attainment of stabilized effective pulmonary ventilation; 4 weeks after the day of attainment of stabilized effective pulmonary ventilation; 3 months after the attainment of stabilized effective pulmonary ventilation
  Neuropsychological test: Preliminary Neuropsychological Battery
Evaluation of cognitive performance: attention and memory - 2 | Baseline (initial visit); day of attainment of stabilized effective pulmonary ventilation; 4 weeks after the day of attainment of stabilized effective pulmonary ventilation; 3 months after the attainment of stabilized effective pulmonary ventilation
  Neuropsychological test: Verbal Span
Evaluation of cognitive performance: attention and memory - 3 | Baseline (initial visit); day of attainment of stabilized effective pulmonary ventilation; 4 weeks after the day of attainment of stabilized effective pulmonary ventilation; 3 months after the attainment of stabilized effective pulmonary ventilation
  Neuropsychological test: Immediate Visual Memory
Evaluation of cognitive performance: attention and memory - 4 | Baseline (initial visit); day of attainment of stabilized effective pulmonary ventilation; 4 weeks after the day of attainment of stabilized effective pulmonary ventilation; 3 months after the attainment of stabilized effective pulmonary ventilation
  Neuropsychological test: Digit Symbol Substitution test
Evaluation of cognitive performance: logical and executive functions - 1 | Day of attainment of stabilized effective pulmonary ventilation; 4 weeks after the day of attainment of stabilized effective pulmonary ventilation; 3 months after the day of attainment of stabilized effective pulmonary ventilation
  Neuropsychological test: Verbal Fluency
Evaluation of cognitive performance: logical and executive functions - 2 | Day of attainment of stabilized effective pulmonary ventilation; 4 weeks after the day of attainment of stabilized effective pulmonary ventilation; 3 months after the day of attainment of stabilized effective pulmonary ventilation
  Neuropsychological test: Progressive Matrices
Evaluation of cognitive performance: logical and executive functions - 3 | Day of attainment of stabilized effective pulmonary ventilation; 4 weeks after the day of attainment of stabilized effective pulmonary ventilation; 3 months after the day of attainment of stabilized effective pulmonary ventilation
  Neuropsychological test: Verbal Analogies
Evaluation of cognitive performance: social cognition | 3 months after the day of attainment of stabilized effective pulmonary ventilation
  Neuropsychological test: Eyes Test
Costs of the T-PEP and IPV treatments - 1 | Through the whole period of clearance treatment to attain a stabilized effective pulmonary ventilation (whole period length is 2 weeks on average)
  Average costs of equipments used in the overall number of sessions with T-PEP or IPV treatments, needed to attain stabilized effective pulmonary ventilation
Costs of the T-PEP and IPV treatments - 2 | Through the whole period of clearance treatment to attain a stabilized effective pulmonary ventilation (whole period length is 2 weeks on average)
  Average costs of consumables used in the overall number of sessions with T-PEP or IPV treatments, needed to attain stabilized effective pulmonary ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Carlotta Stopazzoni, MD, Principal Investigator — Montecatone Rehanilitation Institute SpA
Locations (1):
- Montecatone Rehabilitation Institute S.p.A., Imola, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided